CLINICAL TRIAL: NCT05285280
Title: Prevalence and Risk Factors Associated With Cardiovascular Comorbidity in Men With Erectile Dysfunction
Brief Title: Echocardiography in Men With Erectile Dysfunction
Status: Active, not recruiting | Type: Observational
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Emil Durukan, Principal Investigator, Herlev and Gentofte Hospital
Other Study IDs: EDcard
Record Dates: First submitted 2022-02-02; First posted 2022-03-17 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Erectile Dysfunction; Cardiovascular Diseases; Cardiac Disease
Keywords: Echocardiography; 3D Echocardiography; Strain Rate Imaging; Tissue Doppler; Speckle Tracking
MeSH Terms: conditions — Erectile Dysfunction; Cardiovascular Diseases; Heart Diseases | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echocardiography — The echocardiography will be performed with a GE Vingmed Ultrasoundís Vivid9 (Horten, Norway). All subjects are examined with color TDI, 2-dimensional and M-mode echocardiography, conventional spectral Doppler, 2DSTE, and where possible 4D Echocardiography in the left lateral decubitus position.

SUMMARY:
Cardiovascular disease is the leading cause of morbidity and mortality in the world. To curb disease development, there is, therefore, a need to identify more people at increased risk. This can be done by advanced echocardiography, where the exact contraction pattern and dimensions of the heart are measured.

One group of patients who are already considered to be at increased risk for later development of heart disease are men with erectile dysfunction.

The investigators goal is to study the early detection of cardiac dysfunction in men with erectile dysfunction using both conventional and advanced echocardiography to analyze the possibility of preventing serious cardiovascular disease.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of morbidity and mortality across the globe. About 524,000 Danes live with cardiovascular disease and it affects approx. 56,400 people. In addition, many people live with heart problems without knowing it. These figures emphasize the importance of early identification of more people at increased risk of developing cardiovascular disease to prevent morbidity and mortality.

This can be done using advanced echocardiography, where the heart's precise contraction pattern, as well as structure and dimensions, are measured. One group of patients who are already considered to be at increased risk for later development of cardiovascular disease are men with erectile dysfunction (ED). ED is defined as the persistent inability to achieve or maintain an erection sufficient for satisfactory sexual performance. Approximately 30% of men over the age of 40 are affected by ED, and the incidence increases with age. ED is thought to be a precursor to cardiovascular disease, where it has been proven that after the onset of erection problems, over 3-5 years, there is an approximately 50% increased risk of cardiovascular disease.

The investigators hypothesize that cardiac structure and function assessed by conventional and advanced echocardiography together with cardiac biomarkers are abnormal in patients diagnosed with erectile dysfunction and can identify patients at high risk for cardiovascular complications. Echocardiography can serve as an important tool in risk assessment in these men who do not necessarily have symptom-causing problems.

ELIGIBILITY:
Inclusion Criteria:

* Men above 40 years old diagnosed with ED will be eligible to participate if none of the exclusion criteria below are present.

Exclusion Criteria:

* Patients not able to cooperate
* Patients unable to understand and sign "informed consent"
* Previous pelvic surgery (including prostatectomy, cystectomy and rectal surgery)
* Neurological diseases (e.g. multiple sclerosis, spinal cord injury)
* ED following pelvic trauma

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be invited from the Urology outpatient clinic at Gentofte Hospital.
Sampling Method: Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2032-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of reported cardiac arrest through medical records | 1 year
Number of reported cardiac arrest through medical records | 5 years
Number of reported cardiac arrest through medical records | 10 years
Number of reported hospital admission with heart failure through medical records | 1 year
Number of reported hospital admission with heart failure through medical records | 5 years
Number of reported hospital admission with heart failure through medical records | 10 years
Number of reported peripheral artery disease through medical records | 1 year
  Registration of: Cholesterol levels, blood pressure, claudication and ankle brachial index (ABI).
Number of reported peripheral artery disease through medical records | 5 years
  Registration of: Cholesterol levels, blood pressure, claudication and ankle brachial index (ABI).
Number of reported peripheral artery disease through medical records | 10 years
  Registration of: Cholesterol levels, blood pressure, claudication and ankle brachial index (ABI).
Number of reported coronary heart disease through medical records | 1 year
  Registration of: Coronary angiography
Number of reported coronary heart disease through medical records | 5 years
  Registration of: Coronary angiography
Number of reported coronary heart disease through medical records | 10 years
  Registration of: Coronary angiography
Number of reported hospital admission with acute myocardial infarction through medical records | 1 year
Number of reported hospital admission with acute myocardial infarction through medical records | 5 years
Number of reported hospital admission with acute myocardial infarction through medical records | 10 years
Number of reported angina pectoris through medical records | 1 year
Number of reported angina pectoris through medical records | 5 years
Number of reported angina pectoris through medical records | 10 years
Number of reported ischemic heart disease through medical records | 1 year
Number of reported ischemic heart disease through medical records | 5 years
Number of reported ischemic heart disease through medical records | 10 years

SECONDARY OUTCOMES:
Number of reported all cause mortality | 1 year
Number of reported all cause mortality | 5 years
Number of reported all cause mortality | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Urological Research Unit, Herlev, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No